CLINICAL TRIAL: NCT06189885
Title: Preoperative Daptomycin Prophylaxis for Preventing Gram-Positive or Methicillin-Resistant Staphylococcus Aureus Infection in Two-Stage Exchange Arthroplasty: A Prospective, Randomized, Double-Blinded Trial
Brief Title: Preoperative Daptomycin Prophylaxis in Two-Stage Exchange Arthroplasty: A Prospective, Randomized, Double-Blinded Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 202301864A3
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-11

CONDITIONS: Periprosthetic Joint Infection
MeSH Terms: interventions — Cefazolin; Daptomycin; Vancomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preoperative Daptomycin Prophylaxis in Two-Stage Exchange Arthroplasty (Experimental)
  Interventions: Drug: Cefazolin with Daptomycin
- Preoperative Vancomycin Prophylaxis in Two-Stage Exchange Arthroplasty (Experimental)
  Interventions: Drug: Cefazolin with vancomycin

INTERVENTIONS:
Drug: Cefazolin with Daptomycin — For patients randomized to receive daptomycin (8 mg/kg), the drug will be administered in a 50 cc bag, accompanied by a 500 cc bag of normal saline within 60 minutes before surgical incision and discontinued after 24 hours postoperatively.
  Arms: Preoperative Daptomycin Prophylaxis in Two-Stage Exchange Arthroplasty
Drug: Cefazolin with vancomycin — Then vancomycin (15 mg/kg) will concurrently be given and completed within 60 minutes before surgical incision and discontinued after 24 hours postoperatively9. Patients in the vancomycin arm will receive this drug in a 50 cc bag accompanied by a 500 cc bag of normal saline.
  Arms: Preoperative Vancomycin Prophylaxis in Two-Stage Exchange Arthroplasty

SUMMARY:
The gold standard for treating prosthetic joint infection (PJI) is two-stage exchange arthroplasty. This includes the first stage of debridement and removal of the artificial joint, and the second stage of reimplantation of the artificial joint. Methicillin-resistant staphylococcus aureus (MRSA) infection is one of the factors leading to the failure of artificial joint infection treatment. Before the second stage of the joint surgery, the surgeon will prescribe prophylactic antibiotics based on previous bacterial cultures. The usual preoperative antibiotic is a first-generation cephalosporin antibiotic. If it is MRSA, vancomycin will be given. Increasingly, literature reports link prosthetic joint infections to MRSA, but no changes have been made to the routine recommendation for MRSA prophylactic antibiotic use.

Daptomycin is a cyclic lipopeptide antibiotic that can rapidly penetrate biofilms and bones, and its safety and tolerability have been confirmed. Therefore, it can effectively combat Gram-positive organisms, including MRSA. Daptomycin has many characteristics of an ideal prophylactic: short infusion time, low adverse events during administration, and a range limited to Gram-positive organisms. We aim to assess whether adding antibiotics that cover MRSA would reduce prosthetic joint infections and increase surgical success rates, in addition to the standard recommended prophylactic antibiotics. Thus, this prospective randomized trial is designed to assess, besides using the first-generation cephalosporin antibiotic, the effects of adding an antibiotic with MRSA coverage (Daptomycin vs. Vancomycin).

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 or older with an infection that meets the 2018 International Consensus Meeting (ICM) criteria7 at the time of the first-stage resection arthroplasty with a gram-positive organism, especially MRSA.
2. Will undergo a second stage of reimplantation.

Exclusion Criteria:

1. Patients with a fungal infection or culture-negative infections
2. Known allergies to Cefazolin, Daptomycin, or Vancomycin.
3. Currently receiving surgical treatment for acute postoperative or acute hematogenous PJI.
4. Chronic kidney disease (Creatinine Clearance Rate [CCR] < 30 ml/min/1.73m2)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Infection | One year
  Infection that meets the 2018 ICM criteria after second stage reimplantation.

SECONDARY OUTCOMES:
Acute Kidney Injury | 48 hours
  efined by the Kidney Disease Improving Global Outcomes (KDIGO)11, which includes a rise in serum creatinine by ≥0.3 mg/dl within 48 hours; or an increase in serum creatine ≥1.5 times the patient's preoperative baseline within 7 days; or urine volume <0.5 ml/kg/h for 6 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan